CLINICAL TRIAL: NCT06755255
Title: Evaluation of the Relationship Between Mediterranean Diet and Menopausal Symptoms in Postmenopausal Women Aged 45-56
Brief Title: Evaluation of the Relationship Between Mediterranean Diet and Menopausal Symptoms in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hatice Elif Ozkan Yalcinkaya, Family Medicine Resident, Marmara University Pendik Training and Research Hospital
Other Study IDs: 09.2023.1767
Record Dates: First submitted 2024-11-19; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-11

CONDITIONS: Menopausal Complaints
Keywords: Menopausal Complaints; climacteric; menopausal symptoms; mediterranean diet

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- postmenopausal women aged 45-65: Women who were registered at Tuzla E-ASM affiliated with Marmara University Pendik Hospital and who had been in menopause for at least 1 year

SUMMARY:
This cross-sectional study aimed to evaluate the relationship between the frequency and severity of postmenopausal symptoms in women aged 45-65 years and the level of compliance with the Mediterranean diet, and the main question it aimed to answer is: Do women with higher compliance with the Mediterranean diet have milder symptoms?

DETAILED DESCRIPTION:
This cross-sectional study was conducted between 01.01.2024 and 01.06.2024 with women aged 45-65 who were registered at Tuzla E-ASM affiliated with Marmara University Pendik Hospital and who had been in menopause for at least 1 year. The sample size was calculated as 272 and the target number was determined as 305. After obtaining written consent from the participants who agreed to participate in the study and met the inclusion criteria, a questionnaire form was applied to these individuals, which questioned their sociodemographic characteristics, age of menstruation onset, pregnancy history, smoking and alcohol use, use of supplements, Mediterranean Diet Adherence Scale (MEDAS) and Menopause Rating Scale (MRS). The presence, type and severity of menopausal symptoms with the Mediterranean diet were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Those who volunteered to participate in the study,

Exclusion Criteria:

* Those with a diagnosed eating disorder,
* Those using medication for obesity,
* Those with a chronic metabolic disease that is not receiving treatment and whose values related to the disease are not regulated (pronounced hypo/hyperthyroidism, uncontrolled diabetes, etc.),
* Those with a mental or physical condition that prevents communication (some neuropsychiatric diseases and mental retardation),
* Those who do not understand and/or speak Turkish,
* Those who do not give consent to participate in the study, •-Those who are currently using any hormonal supplements to prevent or reduce menopausal symptoms were excluded from the study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study enrolls only biological females
Study Population: The population of the study consists of all postmenopausal women between the ages of 45-65 registered to Tuzla E-ASM.
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Mediterranean diet adherence and menopausal symptoms association | Data collected at a single time point upon participants' enrollment.
  Mediterranean diet adherence total score and menopausal rating scale total score were inversely and weakly correlated with each other (p<0.01; r= -0.295).

SECONDARY OUTCOMES:
Menopausal symptom severity in women with low and dietary adherence | Data collected at a single time point upon participants' enrollment.
  Women with mild menopausal symptoms had the highest adherence score with the Mediterranean diet, while women with severe symptoms had the lowest adherence score to the Mediterranean diet (p<0.01).
Vasomotor menopausal symptom severity in women with low dietary compliance | Data collected at a single time point upon participants' enrollment.
  Mediterranean diet adherence scores were lower in the group with severe vasomotor symptoms. (p<0,05)
Psychological menopausal symptom severity in women with low dietary compliance | Data collected at a single time point upon participants' enrollment.
  Mediterranean diet adherence scores were lower in the group with severe psychological symptoms.
Urogenital menopausal symptom severity in women with low dietary compliance | Data collected at a single time point upon participants' enrollment.
  There is no significant relationship between urogenital symptom scores and Mediterranean diet compliance scores.

CONTACTS AND LOCATIONS:
Overall Officials: Buğu Usanma Koban, Assistant Professor, Study Director — Marmara University Pendik Training and Research Hospital
Locations (1):
- Marmara University- Tuzla Eğitim ASM, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participant's survey forms
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months
Access Criteria: Forms will only be shared with researchers via Drive

REFERENCES:
- [Background] Ö. Can Gürkan and M. A. Hemşirelik Yüksekokulu Kadın Sağlığı ve Hastalıkları Hemşireliği Araştırma Görevlisi, "MENOPOZ SEMPTOMLARI DEĞERLENDİRME ÖLÇEĞİNİN TÜRKÇE FORMUNUN GÜVENİRLİK VE GEÇERLİLİĞİ."
- [Background] E. Fatma et al., "Turkish Validation and Reliability of Mediterranean Diet Adherence Screener," Pehlivanoglu Ozkan EF. Balcioglu H. Unluoglu I, vol. 42, no. 2, pp. 160-164, 2020, doi: 10.20515/otd.
- [Background] Byrne-Kirk M, Mantzioris E, Scannell N, Villani A. Adherence to a Mediterranean-style diet and severity of menopausal symptoms in perimenopausal and menopausal women from Australia: a cross-sectional analysis. Eur J Nutr. 2024 Oct;63(7):2743-2751. doi: 10.1007/s00394-024-03462-3. Epub 2024 Jul 18. PMID 39026104
- [Background] Herber-Gast GC, Mishra GD. Fruit, Mediterranean-style, and high-fat and -sugar diets are associated with the risk of night sweats and hot flushes in midlife: results from a prospective cohort study. Am J Clin Nutr. 2013 May;97(5):1092-9. doi: 10.3945/ajcn.112.049965. Epub 2013 Apr 3. PMID 23553160
- [Background] Vetrani C, Barrea L, Rispoli R, Verde L, De Alteriis G, Docimo A, Auriemma RS, Colao A, Savastano S, Muscogiuri G. Mediterranean Diet: What Are the Consequences for Menopause? Front Endocrinol (Lausanne). 2022 Apr 25;13:886824. doi: 10.3389/fendo.2022.886824. eCollection 2022. PMID 35546996
- [Background] L. Barrea, G. Pugliese, D. Laudisio, S. Savastano, A. Colao, and G. Muscogiuri, "Does Mediterranean diet could have a role on age at menopause and in the management of vasomotor menopausal symptoms? The viewpoint of the endocrinological nutritionist," 2021. doi: 10.1016/j.cofs.2021.02.018.